CLINICAL TRIAL: NCT02844452
Title: Antipruritic Effect of Acupuncture in Patients With Atopic Dermatitis: Feasibility Study Protocol for a Randomised, Sham-Controlled Trial.
Brief Title: Antipruritic Effect of Acupuncture in Patients With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University (Other)
Responsible Party: Principal Investigator, Kyuseok Kim, assistant professor, Kyunghee University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KOMCIRB-160212-HRBR-004
Record Dates: First submitted 2016-07-15; First posted 2016-07-26 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; acupuncture; visit frequency; adult patient with AD
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Verum Acupuncture 1 (Experimental): The participants with atopic dermatitis in the acupuncture group 1 will attend twelve acupuncture sessions over 4 weeks: 3 days a week. Once the 4-week treatment period was ended, the additional follow-up period will be conducted. The subjects will stand a final visit 4 weeks from the end of treatment period. Any other intervention will not be allowed during this study period.
  Interventions: Device: Acupuncture
- Verum Acupuncture 2 (Experimental): The participants with atopic dermatitis in the acupuncture group 2 will attend eight acupuncture sessions over 4 weeks: 2 days a week. Once the 4-week treatment period was ended, the additional follow-up period will be conducted. The subjects will stand a final visit 4 weeks from the end of treatment period. Any other intervention will not be allowed during this study period.
  Interventions: Device: Acupuncture
- Sham Acupuncture (Sham Comparator): The participants in the sham acupuncture group will visit eight acupuncture sessions over 4 weeks. The acupuncture treatment will be conducted on six control points. The acupressure will be applied with ring-sham press tack needles on three control points. Unlike the acupuncture group 2, partially-individualized manual acupuncture according to the patient's symptoms will not be given but the questions about symptoms will be questioned to patients.
  Interventions: Device: Sham Acupuncture
- Healthy Control (No Intervention): The participants will go through the screening test. The included subjects will complete questionnaires and their blood sample will be obtained.

INTERVENTIONS:
Device: Acupuncture — Acupuncture is a form of alternative medicine and a key component of traditional Korean medicine (TKM) involving thin needles inserted into the body at acupuncture points. It can be associated with the application of heat, pressure, or laser light to these same points. Acupuncture is commonly used for pain relief, though it is also used for a wide range of other conditions. Clinical practice varies depending on the country.
  Arms: Verum Acupuncture 1; Verum Acupuncture 2
Device: Sham Acupuncture — Sham acupuncture is used as a control in scientific studies that test the efficacy of acupuncture in the treatment of various illness or disorders. In an ideal controlled study, subjects would not know whether they were getting true or sham acupuncture. We are going to use Park Sham Acupuncture, which is composed of sham acupuncture needle not penetrating the skin of subjects and Park sham acupuncture device attacted on the subject's skin in order to block the seeing whether the acupuncture needle penetrates skin or not.
  Arms: Sham Acupuncture

SUMMARY:
Introduction: Atopic dermatitis (AD) is a chronic relapsing inflammatory skin disease inducing poor quality of life. Its conventional treatments often cause unsatisfactory relief and adverse effects in long-term application. Acupuncture treatment is regarded to have a curative effect on AD symptoms. The aim of this trial is to evaluate the therapeutic effects of acupuncture on AD symptoms including pruritus and poor quality of life in patients with AD.

Method and Analysis: This trial is a randomized, sham-controlled pilot trial with different visit frequencies. 30 eligible patients with atopic dermatitis will be randomly allocated in a ratio of 1:1:1 to the Verum Acupuncture group 1 (VA1, 3 days weekly), Verum Acupuncture group 2 (VA2, 2 days weekly) and Sham Acupuncture group (2 days weekly). The acupuncture treatment will be given three or two times a week for 4 weeks according to the allocated groups. The main outcome measures are Visual analogue scale for itch (itch VAS), SCORing Atopic Dermatitis (SCORAD) and Eczema Area and Severity Index (EASI) to evaluate the improvement of AD symptoms and Patient Oriented Eczema Measure (POEM), Dermatology Life Quality Index (DLQI) to assess the quality of life of AD patients. It will be measured at baseline, once a week during treatment period and after follow-up period.

Ethics/Dissemination: This protocol was approved by the Institutional Review Boards at Kyung Hee University Korean Medicine Hospital on May 2016. The permission number is KOMCIRB-160212-HRBR-004. This trial will provide the data of therapeutic effects of treating atopic dermatitis with acupuncture in accordance with the different visit frequencies. The outcomes will be facilitated to calculate the sample size of further study with the same design of this study. The findings from this trial will be published and presented in conference.

DETAILED DESCRIPTION:
Objectives This pilot study aims to investigate the feasibility of validating the anti-pruritic effectiveness of the sole acupuncture intervention and the efficacy of different frequent treatments of acupuncture, and discovering noble candidates of a specific biomaterial associated with the development of atopic dermatitis. Moreover, the result will be facilitated in calculating the sample size on the further study.

Trial design A randomized, sham-controlled, different intervention frequency trial will be conducted at the Kyung Hee University Korean Medicine Hospital from June to November 2016.

Participants and Recruitment

Recruitment Acquiring consent will be conducted by the investigators with the principle of informed consent which confirms participants' voluntarism. The participants will sign the document made of general consent form and additional consent provisions for blood collection and use of their human derived material first of all. The exemplary consent paper and other related literature can be offered upon request.

Randomization and allocation concealment The AD patients will be randomized to one of the three groups via block randomization.

An independent statistician will product random numbers with the PROC PLAN of SAS 9.2 (SAS institute Inc., Cary, NC, USA) and transfer them to the Acupuncture and Meridian Science Research Center (AMSRC) at Kyung Hee University where the each randomization number will be sealed in a sequentially numbered non-transparent envelope by a staff uninvolved in this study.

At the beginning of the randomization process, the investigator will call the independent staff in AMSRC to pass the screening number of the participant. Then the AMSRC staff immediately assign the participating patient to one of three groups by unsealing a numbered envelope. It will be documented in the trial master file thoroughly.

Blinding The participating patients and the assessor will be blinded to the group allocation of patients in this trial. It is impossible for acupuncturists to be unaware of the group assignments, but they will not perform the outcome measurements or data analyses.

To prevent a possible bias, the eye patch will be applied for the patients during the acupuncture treatment, and they will be unable to see the practice procedures. All the acupuncture treatment, regardless of the group assignment, will be practiced by using Park sham devices (AcuPrime Co., Ltd., Exeter, UK) which is attached on the applied acupoints as to block the sighting of penetrating or non-penetrating on the skin of acupuncture needles 9. The acupuncture needles and devices will be maintained for 15 min identically.

Intervention Acupuncture treatment Both manual acupuncture treatment and acupressure would be conducted on every participating AD patient. It was designed to become a pragmatic treatment procedure corresponding with real clinic settings.

In this study, the manual acupuncture treatment is composed of basic acupuncture treatment and additional acupuncture treatment: partially individualized acupuncture treatment will be conducted on the basis of the traditional meridian theory and consensus by the experts in acupuncture and the atopic disease. The number of applied acupoints per patient per session ranges from 6 to 19. The optional points include ST43, GB41, LI2, TE3, SI3, TE6, SI2, BL66, LR3 and SP3.

The clinical research coordinator will ask the symptoms associated with additional acupuncture treatment to reduce the bias. The acupuncture treatment will be practiced with a sterilized stainless needle (40 mm length and 0.25 mm diameter; Dongbang Acupuncture Inc., Bundang, Sungnam, Korea) by one same Korean Medicine Docter. Manipulation technique will be performed to elicit 'de qi' sensation. The needle will be inserted in depth of 5 to 30 mm and retained for 15 minute.

Acupressure technique will be taken after the elimination of stainless needles. The 1.5 mm press tack needles (Haeng Lim Seo Won Medical co., China) will be attached on four acupoints per participating patient per session: LI11 bilaterally and auricular-Shenmen contralaterally. It was designed with the traditional meridian theory and consensus by the experts in acupuncture and the atopic disease. The patients will be instructed by the involved staff to press the applied press tack needles located on LI11 when they feel severe pruritus for 3 min.

All the acupuncture practice will be carried out by the same Korean Medicine Doctor, who will be trained for 10 hours to guarantee that he could perform the identical acupuncture treatment according to the pre-constructed protocol.

Dropout criteria on patients' visits During the study period, each patient will visit 12 or 8 treatment sessions according to allocated group. Since frequent visit would be the burden to participating patients and cause absences from the trial, we made the criteria on the absence of participants of each group and the range of dropout. Acupuncture group 1, which have total 12 acupuncture treatment, ought to complete 10 treatment sessions to minimum and acupuncture group 2 and sham acupuncture group, which have total 8 acupuncture treatment, ought to complete 6 sessions. Each treatment session of all the allocated group cannot be delayed over 6 days from the previous session.

Outcome measures One health care provider involved in this study will conduct a series of outcome measures. There will be no separation between primary and secondary outcome since it is an exploratory pilot study to search independent effectiveness of acupuncture intervention on atopic dermatitis and secure a dataset for the further study.

SCORAD index Itch VAS EASI score POEM DLQI CES-D STAXI

Investigating biomaterials with blood collection Serum total IgE measurement Serum cytokine/chemokines measurement Serum cortisol measurement MicroRNA microarray

Statistical Methods Sample size calculation The current trial was established as a pilot study to investigate the anti-pruritic effects of acupuncture for the patients with atopic disease. A total of 30 AD patients, 10 in each group, and 20 healthy controls will be recruited during the study period in regard of 20% dropout rate. Its outcomes will suggest evidences for feasibility of further large-scale study and sample size calculation.

Statistical analysis A statistician uninvolved in the research team will take charge of the statistical analysis by using the SPSS 21.0 (IBM SPSS Statistics, New York, USA). Categorical variables will be provided with percentages and continuous variables will be provided as mean and standard deviation.

The intervention effectiveness will be analyzed with the changes between the baseline and the end of treatment period or follow-up period. Data analysis of baseline characteristics between allocated groups will be compared through a repeated-measures analysis of variance (ANOVA) test and χ2 test respectively on continuous variables and categorical variables.

The different efficiency according to three times or twice weekly acupuncture treatment will be analyzed with the changes in itch VAS and SCORAD index by the Mann-Whitney U-test on continuous variables and χ2 test on categorical variables. The difference on therapeutic efficiency between verum acupuncture treatment groups and sham acupuncture treatment group will be investigated in the same way. And these outcome data will be analyzed with 0.1 (two-sided) statistical significance level and the 90% confidence intervals regarding with the professional advice for the small sample size. For the further study, the difference on treatment groups and control group will be applied to calculate the number of needed participants with a set on 0.05 α and 80% power.

Protection of human subjects Ethical approval and registration This study protocol was approved by the Institutional Review Boards at Kyung Hee University Korean Medicine Hospital (KOMCIRB-160212-HRBR-004). It will be performed in accordance with the standards of the International Committee on Harmonization on Good Clinical Practice and the revised version of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals over age 19
2. Individuals who meet the Hanifin & Rajka and whose AD symptoms express constantly
3. Individuals who check more than 3 points and less than 8 points on the visual analogue scale for atopic dermatitis (with a total score out of 10)
4. Individuals who are graded 10 to 40 points on the SCORAD index
5. Individuals who have not taken the subscribed medicines for atopic dermatitis recent one month.
6. Individuals who understand this study protocol and voluntarily agree with participation.
7. Individuals who have not participated any other researches recent one month

Exclusion Criteria:

1. Individuals whose modalities of atopic dermatitis change unpredictably
2. Individuals who receive inappropriate therapies such as oral corticosteroids which affect the outcomes
3. Individuals who also have asthma, bronchitis or other sever psychological disorders
4. Individuals who have other inappropriate disorders affecting the outcomes

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Itch VAS | Baseline, 1-week, 2-week, 3-week, 4-week, and 8-week
  The itch VAS is one of components of SCORAD index, and it will be particularly applied to assess the severity and alleviation of atopic dermatitis in this trial. The AD patients whose itch VAS scores less than 30 or more than 80 will be excluded because of their lower desire for anti-pruritic therapy or requirement of more potent treatment 13. The change of itch VAS through the trial will be used to classify as responders or non-responders of the acupuncture treatment.
SCORAD index | Baseline, 1-week, 2-week, 3-week, 4-week, and 8-week
  SCORAD is a well-known tool for assessing the severity of atopic dermatitis. The SCORAD contains evaluation of the intensity and extent of affected region and estimation of subjective discomforts, such as pruritus and sleep loss symptom 10-12. SCORAD index contains 6 items to evaluate intensity of atopic dermatitis: erythema, exoriation, edema or papulation, lichenification, oozing or crust, and dryness. The extent of lesion is assessed as percentage of entity. One same KMD will grade the intensity and extent of affected skin and a patient will check their subjective symptoms with visual analogue scale (0 = no itch or sleep loss, 10 = worst imaginable itch or sleep loss).
  The change from baseline SCORAD index at 4 weeks will be analyzed as the primary outcome measure.
EASI score | Baseline, 1-week, 2-week, 3-week, 4-week, and 8-week
  EASI is a validated instrument measuring the severity of atopic dermatitis 12 14. It is composed of distribution of four body regions and four signs of AD: head and neck, trunk, upper extremities, and lower extremities for body regions and erythema, edema/papulation, excoriation, and lichenification for signs of atopic dermatitis. One same KMD will grade the severity of atopic dermatitis with EASI score.
  The change from baseline EASI score at 4 weeks will be analyzed as the primary outcome measure.

SECONDARY OUTCOMES:
POEM | Baseline, 1-week, 2-week, 3-week, 4-week, and 8-week
  POEM is a useful tool for monitoring atopic dermatitis severity which focuses on the patient-reported symptoms and the experienced illness of the patients. Its score ranges 0 to 28 and it is suitable for an outcome measure in the outpatient clinic and in clinical trials 12 15. The participating patient will be introduced to complete the 7-item questionnaire.
DLQI | Baseline, 1-week, 2-week, 3-week, 4-week, and 8-week
  The DLQI is a compact questionnaire which is applicable to patients with any skin disease. It will be reflected to measure the influence of atopic dermatitis on the life of the patient over the previous 7 days. It consists of 10 questions with Likert-type responses and its score ranges from 0 to 30; higher scores imply greater influence on the health-related quality of life .

CONTACTS AND LOCATIONS:
Overall Officials: Kyuseok Kim, PhD, DKM, Principal Investigator — Kyung Hee University Korean Medicine Hospital
Locations (1):
- Kyung Hee University Korean Medicine Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan.

REFERENCES:
- [Derived] Kim YK, Yeom M, Kang S, Park HJ, Kim K, Lee H. Antipruritic Effect of Acupuncture in Patients with Atopic Dermatitis: Feasibility Study Protocol for a Randomised, Sham-Controlled Trial. Evid Based Complement Alternat Med. 2017;2017:1926806. doi: 10.1155/2017/1926806. Epub 2017 Nov 14. PMID 29358961